CLINICAL TRIAL: NCT02686853
Title: Efficacy of Intrathecal Administration of Liposomal Amphotericin B in Cryptococcal Meningitis Without Acquired Immune Deficiency Syndrome
Brief Title: Efficacy of Intrathecal Administration of Liposomal Amphotericin B in Cryptococcal Meningitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hui Bu (Other)
Responsible Party: Sponsor-Investigator, Hui Bu, Study Principal Investigator, Hebei Medical University
Organization: Hebei Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH 003
Record Dates: First submitted 2016-01-26; First posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Cryptococcal Meningitis
Keywords: Intrathecal administration; Liposomal amphotericin B; Without Acquired Immune Deficiency Syndrome
MeSH Terms: conditions — Meningitis, Cryptococcal | interventions — liposomal amphotericin B

ARMS (1):
- Intrathecal administration group (Experimental)
  Interventions: Drug: Liposomal amphotericin B

INTERVENTIONS:
Drug: Liposomal amphotericin B

SUMMARY:
The main purpose of this study is to observe the clinical effect of intrathecal administration of liposomal amphotericin B in Cryptococcal Meningitis without Acquired Immune Deficiency Syndrome (AIDS).

ELIGIBILITY:
Inclusion Criteria:

* Cryptococcus neoformans are found in CSF

Exclusion Criteria:

* Patients with serious heart, lung, liver and renal insufficiency.
* Patients who took broad-spectrum antibiotics and corticosteroids for a long-term.
* Patients with AIDS or obvious immunodeficiency.
* Patients with long term dialysis or intravenous catheter.
* Patients with other brain organic disease such as purulent meningitis, intracranial swelling, etc.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
laboratory examination of cerebrospinal fluid | 2 to 4 weeks
  It includes routine test，biochemistry indicators and cytology ，namely white blood cell count per litre， protein（in g/l），glucose（in mmol/l）and chloride（in mmol/l）in cerebrospinal fluid ，an assessment will be assessed every week

SECONDARY OUTCOMES:
changes of clinical symptoms | 2 to 4 weeks
  headache duration, duration of fever,presence of cranial nerve damage

OTHER OUTCOMES:
The incidence of adverse reactions | 24 hours
  Lower back pain，lower extremity weakness， paraplegia，sphincter disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Bu, MD, Principal Investigator — The Second Hospital of Hebei Medical University